CLINICAL TRIAL: NCT03340376
Title: Prospective Randomized Phase II Trial Comparing Doxorubicin Alone Versus Atezolizumab Alone Versus Doxorubicin and Atezolizumab in Recurrent Cervical Cancer
Brief Title: Doxorubicin Alone Versus Atezolizumab Alone Versus Doxorubicin and Atezolizumab in Recurrent Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGOG-cx3
Record Dates: First submitted 2017-04-05; First posted 2017-11-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — atezolizumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- atezolizumab monotherapy (Experimental): A fixed dose of 1200 mg atezolizumab will be administered intravenously on Day 1 of each 21-day cycle until progressive disease
  Interventions: Drug: Atezolizumab
- atezolizumab combined with doxorubicin (Experimental): A fixed dose of 1200 mg atezolizumab will be administered intravenously on Day 1 of each 21-day cycle. Doxorubicin will be administered on Day 1 of each 21-day cycle at a dose of 75mg/m² for a total of 6 cycles or until progressive disease
  Interventions: Drug: Atezolizumab; Drug: Doxorubicin
- doxorubicin monotherapy (Active Comparator): Doxorubicin will be administered on Day 1 of each 21-day cycle at a dose of 75mg/m² for a total of 6 cycles or until progressive disease
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Atezolizumab — atezolizumab
  Arms: atezolizumab combined with doxorubicin; atezolizumab monotherapy
Drug: Doxorubicin — Doxorubicin
  Arms: atezolizumab combined with doxorubicin; doxorubicin monotherapy

SUMMARY:
This is an open-label, multicenter, randomized phase II trial to evaluate the safety and efficacy of atezolizumab in patients with recurrent cervical cancer in second line therapy. A total of 48 patients will be randomized in 3 arms, each arm consisting of 16 patients:

Arm A: atezolizumab monotherapy q3w Arm B: atezolizumab combined with doxorubicin q3w Arm C: doxorubicin monotherapy q3w

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell or adenocarcinoma of the cervix
* At least one prior chemotherapy regimen for recurrent or advanced disease with a platinum-taxane combination, but not more than two lines of chemotherapy or targeted therapy in recurrent/advanced setting
* Measurable disease
* ECOG≤2
* Adequate pretreatment hematologic, renal and hepatic function test
* Patients are allowed to have had bevacizumab during their prior treatment
* Evidence of non-childbearing status for women of childbearing potential

Exclusion Criteria:

* History of invasive malignancy other than cervical cancer unless there is no recurrence of these other primary tumors the last 3 years.
* Previous anthracycline-based chemotherapy
* Central nerve system metastases and leptomeningeal disease
* Active or history of autoimmune disease
* Prior allogenic bone marrow transplantation or prior solid organ transplantation
* History of idiopathic pulmonary fibrosis
* Known positive test for HIV, or active hepatitis B or hepatitis C
* Known active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Prior immunotherapy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | after 9 months
  after 9 months in the different arms by RECIST v1.1-criteria (doxorubicin, Atezolizumab and the combination of both)

SECONDARY OUTCOMES:
Overall survival | after 24 months
  Overall survival in the different arms (doxorubicin, Atezolizumab and the combination of both)

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Vergote, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No